CLINICAL TRIAL: NCT05953285
Title: The Impact of Sleep Restriction on Gastric Emptying, Appetite and Energy Intake in Healthy Individuals
Brief Title: The Impact of Sleep Restriction on Gastric Emptying, Appetite and Energy Intake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NorthumbiaU
Record Dates: First submitted 2023-03-14; First posted 2023-07-20 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Obesity
Keywords: Sleep restriction; Gastrointestinal function; Appetite regulation; Gut hormones; Hedonic appetite
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The study is a within-subjects, randomized crossover experimental design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted sleep on blood markers and subjective markers of homeostatic, and hedonic appetite (Experimental): The proposed study will take the form of a within-subjects, randomized crossover experimental design. The data will be quantitative. The study will take place for total of approximately 5 weeks / 37 days (+ up to 6 weeks depending on their schedule: Minimum duration = 5 weeks (37 days), Maximum duration = Approximately 11 weeks (79 days).
  Interventions: Other: Sleep restriction
- Restricted sleep on gastric emptying (Experimental): The proposed study will take the form of a within-subjects, randomized crossover experimental design. The data will be quantitative. The study will take place for total of approximately 5 weeks / 37 days (+ up to 6 weeks depending on their schedule: Minimum duration = 5 weeks (37 days), Maximum duration = Approximately 11 weeks (79 days).
  Interventions: Other: Sleep restriction

INTERVENTIONS:
Other: Sleep restriction — The proposed study will take the form of a within-subjects, randomized crossover experimental design. The data will be quantitative.

SUMMARY:
This study aims to examine if partial sleep deprivation results in alterations blood markers and subjective markers of homeostatic, and hedonic appetite, as well as provide initial data as to the impact of sleep restriction on gastric emptying.

DETAILED DESCRIPTION:
The proposed study will take the form of a within-subjects, randomised crossover experimental design. The data will be quantitative. The study will take place for total of approximately 5 weeks / 37 days (+ up to 6 weeks depending on their schedule: Minimum duration = 5 weeks (37 days), Maximum duration = Approximately 11 weeks (79 days).

Following a telephone screening, participants will be provided with a pre-paid envelope containing secondary screening questionnaires in the form of paper documents. Either by drop-off or post to at their place of residence or place of work. The secondary screening documents are detailed under Inclusion / Exclusion criteria and Secondary screening sub-headings. Participants will then return the filled-out inclusion / exclusion documentation if they still desire to take part in the study, either through the pre-paid envelope, or to be picked up by the research team. A member of the research team will then analyse the participants responses and inform them of their eligibility to take part, via email. Following this, participants will be invited to the lab.

Upon entering the lab, participants will be provided with an informed consent form to sign. Following this, demographic information will be collected (Approximately 45 minutes to an hour): This is detailed under the preliminary data collection sub-heading. During this visit, the participant will also be provided with an actigraphy device in order to measure habitual sleep times for one week. Following this, participants will continue to be wear the actigraphy device for a subsequent week, with participants maintaining habitual duration of time in bed, although with (Potentially) altered bedtime, with 7am wake times, in order to standardise participants to 7am wake times and eliminate any erratic sleeping behaviours leading up to the first experimental trial. Participants will also be provided with a food intake and activity diary. The following visits will take the form of experimental trials (Habitual vs 50% habitual sleep): In which the variables of interest will be tested. Namely, blood markers of appetite, self-reported appetite scores, food preference and craving, heart rate variability, gastric emptying, and energy intake. Participants will not be compensated for taking part in the study but will be reimbursed the cost of travelling to and from the lab.

ELIGIBILITY:
Inclusion

1. Healthy (As assessed with medical screening questionnaire)
2. Self-reported habitual bedtimes between 7 to 9 hours (As assessed with the Pittsburgh sleep quality index)
3. Between the ages of 18 to 45

Exclusion

1. Participants will also be excluded from participation if they are pregnant.
2. Current smokers
3. Excessive alcohol (>2 drinks per day)
4. Excessive caffeine (>300mg per day)
5. Musculoskeletal injury.
6. Shift work during the past 4 weeks
7. Travel across more than one time zones during the past 4 weeks.
8. An indication of having a depressed mood (As assessed by a score on the Centre for Epidemiologic Studies of Depression scale above 16).
9. Moderately or highly physically active, as determined by the International Physical Activity Questionnaire (IPAQ) short form.
10. Excessive daytime sleepiness as measured by the Epworth Sleepiness Scale (Score > 10) (ESS) (Hart et al., 2015).
11. Participants will also be considered ineligible if they achieve a score indicative of narcolepsy or chronic insomnia, as assessed through the Pittsburgh Sleep Quality Index [PSQI] (Score > 5) (Hart et al., 2015).
12. Participants must achieve a score < 50 on the Food Craving Questionnaire-Trait-reduced (FCQ-T-r), which has been shown to discriminated between individuals with and without "food addiction" with high sensitivity (85%) and specificity (93%) (Meule et al., 2014).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-01-17 (Estimated); Study Completion 2024-01-17 (Estimated)

PRIMARY OUTCOMES:
Fasting blood markers: Dopamine, Endocannabinoids, Ghrelin, Leptin, Orexin, and Peptide tyrosine tyrosine | Comparisons in fasting blood markers will be made between sleep restricted vs control conditions. A fasted blood sample will be collected during the 5 minute period from 08:10 - 08:15
  A fasting blood sample will be collected in EDTA and Heparin vacutainers in order to assess blood markers of appetite, gastrointestinal function and motivation to feed.
Difference in postprandial blood markers: Dopamine, Endocannabinoids, Ghrelin, Leptin, Orexin, and Peptide tyrosine tyrosine for a breakfast meal | Following the ingestion of a breakfast meal at 08:15, blood will be drawn every 15 minutes until 1 hour postprandially, then every 30 minutes until 3 hours postprandially.
  8 blood sample will be collected in EDTA and Heparin vacutainers in order to assess blood markers of appetite, gastrointestinal function and motivation to feed. Comparisons will be made between sleep restricted vs control conditions for the area under curve (AUC) for the 3 hour postprandial period.
Difference in postprandial blood markers: Dopamine, Endocannabinoids, Ghrelin, Leptin, Orexin, and Peptide tyrosine tyrosine for a lunch-time meal | Following the ingestion of a lunchtime meal at 12:30, blood will be drawn every 15 minutes until 1 hour postprandially, then every 30 minutes until 3 hours postprandially.
  8 blood sample will be collected in EDTA and Heparin vacutainers in order to assess blood markers of appetite, gastrointestinal function and motivation to feed. Comparisons will be made between sleep restricted vs control conditions for the area under curve (AUC) for the 3 hour postprandial period.
Difference in postprandial blood markers: Dopamine, Endocannabinoids, Ghrelin, Leptin, Orexin, and Peptide tyrosine tyrosine for an evening meal | Following the ingestion of an evening meal meal at 16:45, blood will be drawn every 15 minutes until 1 hour postprandially, then every 30 minutes until 3 hours postprandially.
  8 blood sample will be collected in EDTA and Heparin vacutainers in order to assess blood markers of appetite, gastrointestinal function and motivation to feed. Comparisons will be made between sleep restricted vs control conditions for the area under curve (AUC) for the 3 hour postprandial period.
Difference in diurnal blood markers: Dopamine, Endocannabinoids, Ghrelin, Leptin, Orexin, and Peptide tyrosine tyrosine | Blood samples will be drawn at 08:10, and continue to be drawn at regular intervals of 15, 30 and 60 minutes until 20:00.
  27 blood samples will be collected in EDTA and Heparin vacutainers throughout the day, in order to assess blood markers of appetite, gastrointestinal function and motivation to feed. Comparisons will be made between the area under curve (AUC) for the entire diurnal period (11.45 hours), for the sleep restricted vs control conditions.

SECONDARY OUTCOMES:
Difference in gastric emptying of an evening meal | Every 15 mins for 2 hours following test meal. Comparisons will be made between sleep restricted and control conditions.
  Gastric emptying will be measured using the 13-C sodium acetate breath test method Following 2 nights of prescribed sleep of each protocol: Baseline expiratory breath sample will be collected immediately prior to the evening meal of the day then at 15 min intervals post-meal ingestion, for 2 h. This meal will contain 100mg of 13-C Sodium acetate. Expired breath samples will be collected in reusable foil bags using clean, sterilised mouth pieces. Breath samples will be analysed for the ratio of 13CO2:12CO2 by non-dispersive infra-red spectroscopy. The difference in the ratio of 13CO2:12CO2 from baseline breath to post-ingestion breath samples will be expressed as delta over baseline (DOB). Half-emptying time (T½) and time of maximum emptying rate (Tlag) will be calculated.
Difference in subjective feelings of appetite in a fasted state | Ratings of fasting subjective appetite will be collected during the 5 minute period elapsed from 08:10 - 08:15. Comparisons will be made between sleep restricted vs control conditions.
  Subjective measures of appetite will be measured through 100mm visual analogue scales (VAS).100 mm visual analogue scales will be used to assess subjective homeostatic appetite, using paper and pen. Participants will be asked to mark on a line how they rate their current level of subjective appetite as it relates to a series of four questions: With 0mm indicating "Not at all" and 100mm indicating "Extremely". The questions will be, (1) "How strong is your feeling of hunger?", (2) "How strong is your feeling of fullness?", (3) "How Strong is your desire to eat?", and (4) "How much food can you eat right now?", designed to assess hunger, fullness, desire to eat, and prospective food consumption.
Difference in subjective feelings of appetite following a breakfast meal | Every 30 minutes up until 3 hours postprandially, following the ingestion of the test meal at 08:15.
  Subjective measures of homeostatic appetite will be measured through 100mm visual analogue scales (VAS).100 mm visual analogue scales will be used to assess subjective appetite, using paper and pen. Participants will be asked to mark on a line how they rate their current level of subjective appetite as it relates to a series of four questions: With 0mm indicating "Not at all" and 100mm indicating "Extremely". The questions will be, (1) "How strong is your feeling of hunger?", (2) "How strong is your feeling of fullness?", (3) "How Strong is your desire to eat?", and (4) "How much food can you eat right now?", designed to assess hunger, fullness, desire to eat, and prospective food consumption. Comparisons will be made between sleep restricted vs control conditions for the area under curve (AUC) for the 3 hour postprandial period.
Difference in subjective feelings of appetite following a lunch time meal | Every 30 minutes up until 3 hours postprandially, following the ingestion of the test meal at 12:30.
  Subjective measures of homeostatic appetite will be measured through 100mm visual analogue scales (VAS).100 mm visual analogue scales will be used to assess subjective homeostatic appetite, using paper and pen. Participants will be asked to mark on a line how they rate their current level of subjective appetite as it relates to a series of four questions: With 0mm indicating "Not at all" and 100mm indicating "Extremely". The questions will be, (1) "How strong is your feeling of hunger?", (2) "How strong is your feeling of fullness?", (3) "How Strong is your desire to eat?", and (4) "How much food can you eat right now?", designed to assess hunger, fullness, desire to eat, and prospective food consumption. Comparisons will be made between sleep restricted vs control conditions for the area under curve (AUC) for the 3 hour postprandial period.
Difference in subjective feelings of appetite following an evening meal | Every 30 minutes up until 3 hours postprandially, following the ingestion of the test meal at 16:45
  Subjective measures of homeostatic appetite will be measured through 100mm visual analogue scales (VAS).100 mm visual analogue scales will be used to assess subjective homeostatic appetite, using paper and pen. Participants will be asked to mark on a line how they rate their current level of subjective appetite as it relates to a series of four questions: With 0mm indicating "Not at all" and 100mm indicating "Extremely". The questions will be, (1) "How strong is your feeling of hunger?", (2) "How strong is your feeling of fullness?", (3) "How Strong is your desire to eat?", and (4) "How much food can you eat right now?", designed to assess hunger, fullness, desire to eat, and prospective food consumption. Comparisons will be made between sleep restricted vs control conditions for the area under curve (AUC) for the 3 hour postprandial period.
Difference in subjective feelings of appetite throughout the diurnal period. | Every 30 mins throughout the 11.45 hour testing period.
  Subjective measures of homeostatic appetite will be measured through 100mm visual analogue scales (VAS).100 mm visual analogue scales will be used to assess subjective homeostatic appetite, using paper and pen. Participants will be asked to mark on a line how they rate their current level of subjective appetite as it relates to a series of four questions: With 0mm indicating "Not at all" and 100mm indicating "Extremely". The questions will be, (1) "How strong is your feeling of hunger?", (2) "How strong is your feeling of fullness?", (3) "How Strong is your desire to eat?", and (4) "How much food can you eat right now?", designed to assess hunger, fullness, desire to eat, and prospective food consumption. Comparisons will be made between sleep restricted vs control conditions for the area under curve (AUC) for the 11.45 hour postprandial period.
Implicit liking and wanting at mid-day: The Leeds food preference questionnaire (LFPQ) | The LFPQ will be given to participants during the 15 minute period elapsed from 12:15 -12:30, immediately prior to being served the lunchtime meal.
  Subjective hedonic appetite will also be measured using the LFPQ, which has been used previously in studies examining hedonic appetite following a sleep restriction intervention (Radcliffe et al., 2021). This is a computerized task that provides measures of explicit 'liking' and 'wanting' of food preference and reward. As well as preference towards high fat vs low fat, and savoury vs sweet. Participants are presented with an array of pictures of food common in the diet. Foods in the array are chosen from a validated database to be either low or high in fat and similar in familiarity, protein content, sweet or non-sweet taste and palatability. Comparisons will be made between sleep restricted and control conditions.
Implicit liking and wanting in the evening: The Leeds food preference questionnaire (LFPQ) | The LFPQ will be given to participants during the 15 minute period elapsed from 19:45 - 20:00, immediately prior leaving the lab.
  Subjective hedonic appetite will also be measured using the Leeds Food Preference Questionnaire (LFPQ), which has been used previously in studies examining hedonic appetite following a sleep restriction intervention (Radcliffe et al., 2021). This is a computerized task that provides measures of explicit 'liking' and 'wanting' of food preference and reward. As well as preference towards high fat vs low fat, and savoury vs sweet. Participants are presented with an array of pictures of food common in the diet. Foods in the array are chosen from a validated database to be either low or high in fat and similar in familiarity, protein content, sweet or non-sweet taste and palatability. Comparisons will be made between sleep restricted and control conditions.
Heart rate variability (HRV) | Heart rate variability (HRV) data will be gathered from 21:00 on day 2 until 20:00 on day 3, using a polar H9 chest strap heart rate monitor. Differences will be examined between control (Habitual sleep) and intervention (50% of hab
  Spectral analysis of HRV will be used to examine changes to the R-R interval, the time elapsed between two successive R-waves of the QRS heartbeat waveform. This will be used as an estimate for sympathovagal balance, by analysing the differences in ratio of low frequency vs high frequency intervals. Vagal activity will be estimated by analysing the overall high frequency power (HF). Inter-beat intervals shorter than 400 msec or longer than 1700 msec will be considered outliers and will be removed prior to analysis. Comparisons will be made Differences between sleep restricted and control conditions.
Fasting food craving: The Food Cravings Questionnaire-State (FCQ-S) | Scores will be gathered in a fasted state during the 5 minute period elapsed from 08:10 - 08:15. Comparisons will be made between sleep restricted vs control conditions.
  The Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items:
  An intense desire to eat (Items 1, 2, 3) Anticipation of positive reinforcement that may result from eating (Items 4, 5, 6) Anticipation of relief from negative states and feelings as a result of eating (Items 7, 8, 9) Lack of control over eating (Items 10, 11, 12) Craving as a physiological state (i.e., hunger) (Items 13, 14, 15). Response categories range from 1 = strongly disagree to 5 = strongly agree.
  This will be provided immediately prior to serving the breakfast meal.
Postprandial food craving, breakfast: The Food Cravings Questionnaire-State (FCQ-S) | Scores will be gathered during the 5 minute period elapsed from 08:30 - 08:35 following the breakfast meal. Comparisons will be made between sleep restricted vs control conditions.
  The Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items:
  An intense desire to eat (Items 1, 2, 3) Anticipation of positive reinforcement that may result from eating (Items 4, 5, 6) Anticipation of relief from negative states and feelings as a result of eating (Items 7, 8, 9) Lack of control over eating (Items 10, 11, 12) Craving as a physiological state (i.e., hunger) (Items 13, 14, 15). Response categories range from 1 = strongly disagree to 5 = strongly agree.
  This will be provided immediately following ingestion of the breakfast meal.
Preprandial food craving, lunch: The Food Cravings Questionnaire-State (FCQ-S) | Scores will be gathered during the 5 minute period elapsed from 12:25 - 12:30, prior to the lunchtime meal. Comparisons will be made between sleep restricted vs control conditions.
  The Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items:
  An intense desire to eat (Items 1, 2, 3) Anticipation of positive reinforcement that may result from eating (Items 4, 5, 6) Anticipation of relief from negative states and feelings as a result of eating (Items 7, 8, 9) Lack of control over eating (Items 10, 11, 12) Craving as a physiological state (i.e., hunger) (Items 13, 14, 15). Response categories range from 1 = strongly disagree to 5 = strongly agree.
  This will be provided immediately prior to serving the lunchtime meal.
Postprandial food craving, lunch: The Food Cravings Questionnaire-State (FCQ-S) | Scores will be gathered during the 5 minute period elapsed from 12:45 - 12:50, following the lunchtime meal. Comparisons will be made between sleep restricted vs control conditions.
  The Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items:
  An intense desire to eat (Items 1, 2, 3) Anticipation of positive reinforcement that may result from eating (Items 4, 5, 6) Anticipation of relief from negative states and feelings as a result of eating (Items 7, 8, 9) Lack of control over eating (Items 10, 11, 12) Craving as a physiological state (i.e., hunger) (Items 13, 14, 15). Response categories range from 1 = strongly disagree to 5 = strongly agree.
  This will be provided immediately following ingestion of the lunchtime meal.
Preprandial food craving, evening meal: The Food Cravings Questionnaire-State (FCQ-S) | Scores will be gathered during the 5 minute period elapsed from 16:40 - 16:45, prior to the evening meal. Comparisons will be made between sleep restricted vs control conditions.
  The Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items:
  An intense desire to eat (Items 1, 2, 3) Anticipation of positive reinforcement that may result from eating (Items 4, 5, 6) Anticipation of relief from negative states and feelings as a result of eating (Items 7, 8, 9) Lack of control over eating (Items 10, 11, 12) Craving as a physiological state (i.e., hunger) (Items 13, 14, 15). Response categories range from 1 = strongly disagree to 5 = strongly agree.
  This will be provided immediately prior to serving the evening meal.
Postprandial food craving, evening meal: The Food Cravings Questionnaire-State (FCQ-S) | Scores will be gathered during the 5 minute period elapsed from 17:00 - 17:05 following the evening meal. Comparisons will be made between sleep restricted vs control conditions.
  The Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items:
  An intense desire to eat (Items 1, 2, 3) Anticipation of positive reinforcement that may result from eating (Items 4, 5, 6) Anticipation of relief from negative states and feelings as a result of eating (Items 7, 8, 9) Lack of control over eating (Items 10, 11, 12) Craving as a physiological state (i.e., hunger) (Items 13, 14, 15). Response categories range from 1 = strongly disagree to 5 = strongly agree.
  This will be provided immediately following ingestion of the evening meal.
Night-time food craving, end of trial: The Food Cravings Questionnaire-State (FCQ-S) | Scores will be gathered during the 5 minute period elapsed from 20:00 - 20:05 immediately prior to leaving the lab. Comparisons will be made between sleep restricted vs control conditions.
  The Food Cravings Questionnaire-State (FCQ-S) measures the intensity of momentary food craving. The questionnaire has 15 items:
  An intense desire to eat (Items 1, 2, 3) Anticipation of positive reinforcement that may result from eating (Items 4, 5, 6) Anticipation of relief from negative states and feelings as a result of eating (Items 7, 8, 9) Lack of control over eating (Items 10, 11, 12) Craving as a physiological state (i.e., hunger) (Items 13, 14, 15). Response categories range from 1 = strongly disagree to 5 = strongly agree.
  This will be provided immediately following ingestion of the evening meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom